CLINICAL TRIAL: NCT03935971
Title: The Effects of Dupilumab on Allergic Contact Dermatitis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ari Goldminz, Instructor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P002882
Record Dates: First submitted 2019-04-23; First posted 2019-05-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with Allergic Contact Dermatitis (Experimental): Dupilumab 600 mg/4 mL subcutaneously once, then 300 mg/2 mL every 2 weeks for 10 weeks
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — See arm/group description

SUMMARY:
The aim of this study is to investigate the effects of dupilumab on allergic contact dermatitis.

DETAILED DESCRIPTION:
The investigators will recruit 30 patients with allergic contact dermatitis who have not improved with allergen avoidance up to 18 months after patch testing, but where allergic contact dermatitis is still suspected. Subjects will receive 10 weeks of dupilumab, and both clinical data and tissue samples will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. At least one contact allergen with a 2+ (strong) or 3+ (extreme reaction) confirmed by patch testing within 6 months of the baseline visit that can be duplicated at the initiation of the study (placement at Week 0 and patch test reaction read at Week 0 +72-120 hours).
3. Allergic contact dermatitis diagnosed clinically by the principle investigators who have expertise in allergic contact dermatitis
4. Investigator's global assessment score of at least 3 (range 0-4) at the screening and baseline visits
5. Documented recent history (within 18 months of patch testing) of inadequate response to treatment with topical medications and allergen avoidance
6. Able and willing to provide informed consent, participate in study visits, and undergo visit procedures

Exclusion Criteria:

1. Prior dupilumab use
2. Treatment with a systemic immune-regulating medication within 3 months of the baseline visit or the patient's prior patch testing, whichever is longer. Examples of these medications include azathioprine, methotrexate, mycophenolate mofetil, Janus kinase inhibitors, and phototherapy (including tanning booths). Cyclosporine or prednisone may not have been used within 1 month of the baseline visit.
3. Treatment with other biologic agents, such as TNF inhibitors, anti-IL 17 agents, anti-IL 12/23 agents, or anti-IL 23 agents, within 4 months of baseline visit or the patient's prior patch testing, whichever is longer.
4. Use of rituximab within at 6 months (or until lymphocyte counts have normalized if longer than 6 months) of the baseline visit or the patient's prior patch testing, whichever is longer.
5. Treatment with topical corticosteroids or topical calcineurin inhibitors within 1 week before the baseline visit
6. Other active conditions, such as psoriasis, that may confound clinical evaluations of dermatitis and patient-reported symptoms
7. Increased risk of infection or reactivated infection, including history of human immunodeficiency virus, hepatitis B, hepatitis C, endoparasitic infections, receipt of a live attenuated vaccine within 3 months of the baseline visit, chronic or acute infection requiring treatment within 4 weeks of the baseline visit, immunosuppressed status (ie recurrent or resistant opportunistic infections)
8. Malignancy within 5 years of the screening visit excluding local cutaneous squamous cell carcinoma, basal cell carcinoma or cervical carcinoma in situ that has been fully treated.
9. Women who are or plan to become pregnant or breastfeed during study participation or are unable or not willing to use birth control during the study and for 4 months after the last dose of dupilumab. Options for birth control include abstinence, double barrier (ie male condom and female diaphragm), vasectomy, intrauterine device, and hormonal contraception. Females who have not had menses within 1 year of the baseline, bilateral tubal ligation, hysterectomy, and/or bilateral oophorectomy visit do not require additional methods contraception during study participation.
10. Unstable condition or status, as per study investigator's judgment, that may lead to more likely discontinuation from the study including but not limited to major, recurrent medical illnesses that may require hospital admission and/or discontinuation of dupilumab, surgery that would require discontinuation of dupilumab and/or major rehabilitation, inability to participate in all study visits and administer dupilumab
11. Resident outside of Massachusetts, Connecticut, Rhode Island, New Hampshire, Maine or Vermont state.
12. Unable to use Zoom videoconferencing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Investigator's Global Assessment (IGA) score | week 0, week 6, week 12
  The investigator's global assessment is a physician-reported global assessment of disease activity (range 0-4) with 0 being clear and 4 being severe

SECONDARY OUTCOMES:
Change in Body Surface Area (BSA) | week 0, week 6, week 12
  The body surface area is a physician-reported measure of the amount of disease involvement. The patient's palm size approximates 1% of body surface area involvement.
Change in Eczema Area and Severity Index (EASI) score | week 0, week 6, week 12
  The eczema-area-and-severity-index score is a composite score of disease severity and extent of disease distribution. It was initially developed for evaluation of eczema. Disease severity (range 0-3; 0 being no disease and 3 being severe disease) is a measure of redness, thickness/induration, scratching, and lichenification. Each characterization is measured separately for body regions (head and neck, trunk, upper extremities, and lower extremities) to calculate a regional score. The total score is a sum of the four body regions (range 0-72).
Change in Numerical Rating Scale (NRS) itch | week 0, week 6, week 12
  The numerical rating scale for itch is a patient-reported measure of itch (range 0-10) with 0 being no itch and 10 being the worst imaginable itch.
Change in Dermatology Life Quality Index (DLQI) | week 0, week 6, week 12
  The Dermatology Life Quality Index is a 10-question, patient-reported instrument to assess impact of skin diseases on patient quality of life.
Change in SLEEPY-Q (Sleep Questionnaire) score | week 0, week 6, week 12
  The Sleepy-Q is a patient-derived, patient-reported sleep questionnaire for patients with chronic inflammatory dermatoses that consists of 28 individual questions. It assesses four dimensions of sleep in patients with inflammatory skin conditions: sleep disturbance (overall score 0-40, 0 being "no sleep disturbance" and 40 being "severe sleep disturbance"), causes of sleep disturbance related to dermatitis (binary, yes/no), causes of sleep disturbance unrelated to dermatitis (binary, yes/no), and impairment related to sleep disturbance (two subscales including Life Impairment Score = overall 0-40, being 0 "no life impairment" and 40 "severe life impairment" and Dermatitis Impairment Score = overall 0-30, being 0 "no impairment" and 30 "severe impairment." The total impairment related to sleep disturbance is scored overall 0-70 after summing of the two subscales).
Skin Samples | week0+72-120 hours and week 12+72-120 hours
  Inflammatory markers (Th1, Th2, Th17, Th22 immune pathways) in the skin of patients will be evaluated before and after dupilumab.
Blood Samples | week 0, week0+72-120 hours, week 12 and week 12+72-120 hours
  Inflammatory markers (Th1, Th2, Th17, Th22 immune pathways) in the blood of patients will be evaluated before and after dupilumab.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Department of Dermatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No